CLINICAL TRIAL: NCT06016998
Title: Prediction Model of Hypoxemia in Gastrointestinal Endoscopy Based on Facial Photography and Clinical Indicators
Brief Title: Prediction Model of Hypoxemia in Gastrointestinal Endoscopy Sedation
Status: Completed | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Mengchang Yang, Deputy Chief Physician, Sichuan Provincial People's Hospital
Other Study IDs: FACIAL-123
Record Dates: First submitted 2023-05-21; First posted 2023-08-30 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Hypoxemia During Surgery
Keywords: Hypoxemia; Sedation; Prediction
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of hypoxemia during gastrointestinal endoscopy sedation is high, but there is still a lack of perfect prediction model of hypoxemia, which often leads to unpredictable respiratory complications. In order to ensure the safety of gastrointestinal endoscopy sedation and make emergency plans in advance, a better diagnostic model is urgently needed to help assess the risk of hypoxemia in patients undergoing the process and make early intervention measures. Facial photography is a simple and feasible measure that can show the facial soft tissue and structure of bone. The purpose of this study is to explore whether facial photography combined with other clinical indicators can build a prediction model of hypoxemia during gastrointestinal endoscopy sedation.

DETAILED DESCRIPTION:
Gastrointestinal endoscopy is an effective method for diagnosing gastrointestinal diseases. There is a increasing number of patients undergo gastrointestinal examinations year by year. Drug sedation can improve patient comfort and increase the intraoperative detection rate of digestive disease. At present, the most commonly used medication for gastrointestinal endoscopy sedation is propofol, which has a fast onset and short duration of time, making it very suitable for sedation during outpatient short surgeries. However, propofol can cause intraoperative hypoxemia. The hypoxemia is mainly caused by the respiratory inhibition of propofol and upper airway obstruction after anesthesia. Hypoxemia caused by respiratory inhibition can be optimized by adjusting the dose regimen. Hypoxemia caused by upper airway collapse is more urgent and more difficult to deal with, and usually requires suspension of gastroscopy and uses mask to ventilation , even needs undergo tracheal intubation. If patients suffer from hypoxemia for a long time, it can lead to myocardial ischemia, arrhythmia, permanent nerve injury, and even death and other serious complications. Conventional airway assessment methods have poor prediction ability for airway abnormalities, and imaging refined measurement indicators have good prediction ability, but their implementation is difficult and difficult to promote. At present, there is still a lack of accurate and simple prediction model for hypoxemia. It is still difficult to make a complete early warning for intraoperative respiratory complications, and intraoperative hypoxemia still occurs frequently. Therefore, in order to ensure the safety of gastrointestinal endoscopy sedation and make emergency plans in advance, a more complete diagnostic model is urgently needed to help assess the risk of hypoxemia in patients undergoing painless gastrointestinal endoscopy surgery and make early interventions.

Based on the above, the investigators assume that facial photography can provide a comprehensive measurement of risk factors for craniofacial bone and soft tissue (obesity). A prediction model constructed by combining facial photography measurement indicators with other relevant indicators can easily and efficiently predict airway abnormalities. Therefore, this study mainly explores the prediction model of craniofacial phenotype based on facial photos and combined clinical indicators for hypoxemia after gastrointestinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Patients undergoing painless gastroscopy
3. The American Society of Anesthesiologists (ASA) grades I to III;
4. The basic oxygenation SPO2 of the patient's breathing indoor air is ≥ 96%

Exclusion Criteria:

1. Have a history of symptomatic craniofacial abnormalities (such as Down syndrome)
2. Previous history of craniofacial surgery
3. There is too much facial hair, which clearly blurs the facial markings.
4. Severe cardiopulmonary diseases such as myocardial infarction and bronchial asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing painless gastroscopy in Sichuan Provincial People's Hospital
Sampling Method: Probability Sample
Enrollment: 1023 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Measurement of facial features | 1 day During the process of anesthesia assessment
  Measuring 50 sets of facial features through 5 facial photos

SECONDARY OUTCOMES:
BMI | 1 day During the process of anesthesia assessment
  Weight and height will be combined to report BMI in kg/m^2
Neck circumference | 1 day During the process of anesthesia assessment
  Measure the neck circumference at the level of cricoid cartilage
waist circumference | 1 day During the process of anesthesia assessment
  Measure waist circumference at navel level
Modified Mallampati Score | 1 day During the process of anesthesia assessment
  The patient is asked to sit upright, with the head in the center, the mouth as wide as possible, the tongue as far out as possible, no pronunciation is required, the pharyngeal structure is observed, and the observation is repeated twice to avoid false positives or false negatives.It is divided into four levels according to the structure of the pharynx.Higher level indicates difficulty in airway management.

OTHER OUTCOMES:
Thyromental Distance | 1 day During the process of anesthesia assessment
  Measure the distance from thyroid cartilage to the chin.If the distance is less than six centimeters, it indicates difficulty in airway management.
Upper lip bite test | 1 day During the process of anesthesia assessment
  The patient is in a sitting position, with the lower jaw extending forward as much as possible and using the lower incisor to bite the lip line of the upper lip as much as possible. The level I lower incisor bites above the lip line of the upper lip; Level II lower incisors can bite below the red lip of the upper lip; Level III lower incisors cannot bite the upper lip.Higher level indicates difficulty in airway management.
interincisor gap | 1 day During the process of anesthesia assessment
  Measure the distance between the upper and lower incisors .If the distance is less than three centimeters, it may indicate difficulty in airway management.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China